CLINICAL TRIAL: NCT07278804
Title: Development of a Pain Control Options Menu for IUD Insertion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00117230
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: IUD Insertion Pain
Keywords: IUD insertion; Pain control options menu; Pain control
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Will initially enroll a control group that does not receive any intervention, after control group data is complete, will enroll for the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No menu - control group (No Intervention): Control group - no intervention administered
- Menu - intervention group (Experimental): Participants will receive the pain control options menu prior to IUD insertion
  Interventions: Other: Pain control options menu

INTERVENTIONS:
Other: Pain control options menu — A menu of pain control options available to participants to choose from during IUD (intrauterine device) insertion procedure
  Arms: Menu - intervention group

SUMMARY:
The goal of this study is to evaluate if using a pain management options menu for IUD (intrauterine device) insertion improves patient autonomy, satisfaction, and/or pain. The main questions it aims to answer are:

Does a pain management options menu for IUD insertion improve patient autonomy? Does a pain management options menu for IUD insertion improve patient satisfaction? Does a pain management options menu for IUD insertion improve patient pain?

Researchers will compare survey data from patients receiving IUDs before and after a pain management options menu is implemented.

Participants will be asked to answer survey questions addressing their feelings of autonomy, satisfaction, and pain in regards to their IUD insertion experience.

DETAILED DESCRIPTION:
The investigators are developing a pain management options menu to be given to patients who are undergoing IUD insertion with the goal of improving patient autonomy, satisfaction, and pain scores. The investigators will give patients a survey exploring these aspects of the IUD insertion experience and compare the survey results from patients who were surveyed before the menu was implemented and after the menu was implemented.

ELIGIBILITY:
Inclusion Criteria:

* Having an IUD placed in a clinic visit
* Able to read and speak English
* Age 18-50 years old

Exclusion Criteria:

* Having an IUD placed in the operating room under general anesthesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Modified PCCC Autonomy Score | Day of study enrollment/IUD insertion
  A modified version of the Person-Centered Contraceptive Care (PCCC) scale will be used to measure patient autonomy. This scale is a 4-item questionnaire evaluating provider performance regarding respect for patients, information provision, and eliciting and honoring patient preferences for birth control. The total score will be a number between 4 and 20.

SECONDARY OUTCOMES:
Highest level of pain experienced | Day of IUD insertion procedure, 24 hours after IUD insertion procedure
  Patients will be asked to rate the highest level of pain that they experienced during IUD insertion/during the 24 hours after IUD insertion on a scale from 0-10.
Number of participants in which pain felt met expectations | Day of IUD insertion procedure, 24 hours after IUD insertion procedure
  Patients will be asked whether the pain they experienced was less than, the same as, or more pain than they expected.
Patient satisfaction score | Day of IUD insertion procedure, 24 hours after IUD insertion procedure
  Patient's will be asked to rate their overall satisfaction with their IUD insertion experience on a scale from 0-10.
Number of participants who would choose an IUD for contraception again | Day of IUD insertion procedure, 24 hours after IUD insertion procedure
  Patient will be asked whether they would choose an IUD for contraception again based on their IUD insertion experience. Answer options will be yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Thomason, MD, MPH, Principal Investigator — Duke University Hospital
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.